CLINICAL TRIAL: NCT06561477
Title: Study of the Validity of Intensive Care Cirrhosis Outcome Score (ICCO) in Predicting Outcome in Cirrhotic Patients Admitted to Intensive Care Unit.
Brief Title: Role of ICCO Score in Predicting Outcome in ICU Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Mamdouh Nathan, principle investigator, Assiut University
Other Study IDs: ICCO score
Record Dates: First submitted 2024-08-09; First posted 2024-08-20 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intensive care cirrhosis outcome (ICCO) score — ICCO score will be calculated for the participants to use it as a predictor for mortality and ICU outcome The ICCO score is 0.3707 + (0.0773 x bilirubin (mg/dl)) - (0.00849 x cholesterol (mg/dl)) -(0.0155 x creatinine clearance (ml/min)) + (0.1351 x lactate (mmol/l))

SUMMARY:
This study aims at calculating a specific score to cirrhotic patients admitted at ICU (ICCO score) and use this score to predict mortality and outcome for admitted patients.

DETAILED DESCRIPTION:
Liver cirrhosis is the final stage of chronic liver disease. It is characterized by an irreversible replacement of liver parenchyma with fibrotic tissue and regenerative nodules. The major causes of cirrhosis include hepatitis B virus and hepatitis C virus infection, alcohol-associated liver disease (ALD), and non-alcoholic fatty liver disease (NAFLD).

The prognosis of cirrhotic patients admitted to the ICU remains poor It was reported that the mortality rate of patients with cirrhosis admitted to an intensive care unit (ICU) due to organ dysfunction ranges from 34% to 69% depending on the cause of admission, the presence of organ failure (OF) and the severity of the underlying liver disease.

Several prognostic scoring systems have been used to assess patients with cirrhosis admitted to the ICU, general ICU mortality risk scores; such as the Sequential Organ Failure Assessment (SOFA) score and the Acute Physiology and Chronic Health Evaluation II (APACHE II) score, other liver specific scores such as Model of end stage liver disease (MELD) score.

These scores can be calculated immediately upon admission to the ICU (first 24 h) or during the first days of hospitalization, leading to an evolutionary assessment over this short period of time.

Intensive care cirrhotic outcome (ICCO) score is a new score that was introduced to predict mortality and ICU outcome in cirrhotic patients admitted to the ICU. with limited studies that test the validity of the score and compare it with the other well-known ICU scores.

In clinical practice, it remains controversial to determine which score is better at predicting overall mortality, this is due to that Each score is calculated according to its own criteria, and only data obtained within the first 24 hours of the first ICU admittance is used.

In this study investigators will test the validity of ICCO score and compare it with other different ICU scores to find out the most useful score in early prediction of ICU outcome for cirrhotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age ≥18 years) with cirrhosis admitted to the ICU.
* Confirmed diagnosis of cirrhosis based on clinical, radiological, and/or histological criteria.
* Need for intensive care management due to acute illness or complications related to cirrhosis.

Exclusion Criteria:

* Patients without a confirmed diagnosis of cirrhosis.
* Patients with acute liver failure not meeting criteria for cirrhosis.
* Patients with incomplete data for calculating ICCO.
* Patients transferred from another ICU.
* Patients who refuse participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with confirmed diagnosis with liver cirrhosis admitted to the intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Testing the validity of ICCO score in predicting mortality in critically ill patients with cirrhosis admitted to the ICU. | baseline
  ICCO score will be calculated to all participants based on the formula The ICCO score was 0.3707 + (0.0773 x bilirubin (mg/dl)) - (0.00849 x cholesterol (mg/dl)) -(0.0155 x creatinine clearance (ml/min)) + (0.1351 x lactate (mmol/l)). and then correlation between ICCO score and ICU mortality will be tested

SECONDARY OUTCOMES:
Compare ICCO score with other established ICU scoring systems regarding their ability to predict mortality in ICU cirrhotic patients. | baseline
  each score of these scores will be calculated to all patients at time of ICU admission, follow up will be done until end of ICU stay, then statistical analysis will be done to compare the effectiveness of each score in prediction of mortality.
Evaluate the utility of ICCO score in guiding clinical decision-making and resource allocation in ICU settings. | baseline
  after statistical analysis of collected data, if the ICCO score has good predictive value, then it can be used to make clinical decision for admission of patients to ICU or not depending of the prediction of their outcomes using the ICCO score.
Assess the correlation of ICCO score with severity of liver disease and other organ dysfunctions. | baseline
  ICCO score value will be calculated to all participants and statistical analysis will be done to find any correlation between ICCO score and degree of severity of liver disease.

REFERENCES:
- [Background] Zauner C, Schneeweiss B, Schneider B, Madl C, Klos H, Kranz A, Ratheiser K, Kramer L, Lenz K. Short-term prognosis in critically ill patients with liver cirrhosis: an evaluation of a new scoring system. Eur J Gastroenterol Hepatol. 2000 May;12(5):517-22. doi: 10.1097/00042737-200012050-00007. PMID 10833094
- [Background] Gumilas NSA, Widodo I, Ratnasari N, Heriyanto DS. Potential relative quantities of miR-122 and miR-150 to differentiate hepatocellular carcinoma from liver cirrhosis. Noncoding RNA Res. 2022 Feb 6;7(1):34-39. doi: 10.1016/j.ncrna.2022.01.004. eCollection 2022 Mar. PMID 35224317
- [Background] Huang DQ, Terrault NA, Tacke F, Gluud LL, Arrese M, Bugianesi E, Loomba R. Global epidemiology of cirrhosis - aetiology, trends and predictions. Nat Rev Gastroenterol Hepatol. 2023 Jun;20(6):388-398. doi: 10.1038/s41575-023-00759-2. Epub 2023 Mar 28. PMID 36977794
- [Background] Abdellatif Z, Eletreby R, Samir R, Abdallah M, Lithy R, Zayed N. Outcome and prognostic markers of cirrhotic and non-cirrhotic patients admitted to a hepatology ICU in a tertiary care university hospital. Afr Health Sci. 2022 Jun;22(2):377-383. doi: 10.4314/ahs.v22i2.43. PMID 36407342
- [Background] da Silveira F, Soares PHR, Marchesan LQ, da Fonseca RSA, Nedel WL. Assessing the prognosis of cirrhotic patients in the intensive care unit: What we know and what we need to know better. World J Hepatol. 2021 Oct 27;13(10):1341-1350. doi: 10.4254/wjh.v13.i10.1341. PMID 34786170
- [Background] Elzouki AN, Suliman S, Alhasan R, Abdullah A, Othman M, Badi A. Predicting mortality of patients with cirrhosis admitted to medical intensive care unit: An experience of a single tertiary center. Arab J Gastroenterol. 2016 Dec;17(4):159-163. doi: 10.1016/j.ajg.2016.11.003. Epub 2016 Dec 15. PMID 27988236
- See also: Related Info — https://zumj.journals.ekb.eg/article_349869.html